CLINICAL TRIAL: NCT01243970
Title: Randomised, Double-blind, Phase IV Study to Compare the Incidence of ECG Changes During Elective Caesarean Section Under Spinal Anaesthesia When Using Phenylephrine or Ephedrine Infusion to Maintain Baseline Systolic Blood Pressure
Brief Title: Ephedrine vs Phenylephrine - ECG Changes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Change in clinical practice since the start of the trial in 2011 (phenylephrine superior)
Sponsor: University College London Hospitals (Other)
Collaborators: Obstetric Anaesthetists' Association United Kingdom (Other)
Responsible Party: Principal Investigator, Roshan Fernando, chief investigator, University College London Hospitals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08/0182
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Spinal Anesthesia; Pregnancy
Keywords: Spinal anaesthesia; phenylephrine; ephedrine; ECG changes; Caesarean delivery; Myocardial ischaemia; Cardiac output; hypotension
MeSH Terms: conditions — Coronary Artery Disease; Hypotension | interventions — Phenylephrine; Ephedrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- phenylephrine infusion (Active Comparator)
  Interventions: Drug: Phenylephrine
- Ephedrine infusion (Active Comparator)
  Interventions: Drug: Ephedrine

INTERVENTIONS:
Drug: Phenylephrine — Infusion dose 50 mcg / minute. On/off regimen in response to blood pressure (BP) readings every minute. Approximative 30 minutes treatment duration. Total dose 50 mcg - 1500 mcg *
  * We will start the infusion after the spinal anaesthetic (see trial design), and while we will monitor cardiac output and BP (for 20 minutes) the surgeons will prep the patient (surgery not started yet). Birth should occur more or less 10-15 minutes after beginning surgery, so this is approximatively 30 minutes after spinal anaesthetic. It is very unlikely that the infusion will run continuously and exceed 1500 mcg.
  Arms: phenylephrine infusion
Drug: Ephedrine — Infusion dose 4mg / minute. On/off regimen in response to blood pressure readings every minute. Approximative 30 minutes treatment duration. Total dose 4 mg - 120 mg. *
  * We will start the infusion after the spinal anaesthetic(see trial design), and while we will monitor cardiac output and BP (for 20 minutes) the surgeons will prep the patient (surgery not started yet). Birth should occur more or less 10-15 minutes after beginning surgery, so this is approximatively 30 minutes after spinal anaesthetic. It is very unlikely that the infusion will run continuously and exceed 120mg.
  Arms: Ephedrine infusion

SUMMARY:
ECG changes during caesarean section are common. Incidence of ST depression on the ECG is up to 81% in some studies. Although this may indicate inadequate oxygen supply to the heart muscle (myocardial ischaemia) many other theories have been suggested including air entering the circulation from the placental bed, high heart rate, hormone or nervous system influences and spasm of the coronary blood supply. Perioperative ST depression often reflects an imbalance between heart muscle oxygen supply and demand. At the time of delivery, high heart rate is common and there is a further increase in the amount of blood the heart has to pump every minute due to blood coming back to the circulation from the placental bed. This increases oxygen demand and most ST changes are seen at the time of delivery or within 30 minutes. The clinical significance of these changes is much debated, and apart from a few case reports do not appear to be associated with poor heart muscle function or ischaemia (lack of oxygen supply). Management of the mother's blood pressure during caesarean section has changed greatly in recent years. Intermittent boluses of ephedrine, given when blood pressure is low, have been replaced with prevention of low blood pressure and phenylephrine has become the drug of choice. Ephedrine increases heart rate and contractility of the heart muscle and is likely to increase oxygen demand. Phenylephrine reduces heart rate while maintaining blood pressure which may result in a more favorable oxygen supply demand ratio.

The investigators aim to compare the incidence of ECG changes if the mother's blood pressure is maintained with phenylephrine as compared to ephedrine. To see if these ECG changes are associated with myocardial ischaemia, the investigators will perform troponin T analysis after delivery. Troponin T is a molecule released by ischaemic heart muscle.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give written informed consent
2. >37/40 weeks gestation
3. Singleton pregnancy
4. Elective caesarean section under spinal anaesthesia
5. In good general health (American Society of Anesthesiology Category 1 or 2, fit and well or with mild systemic disease that has no impact on physical activity )

Exclusion Criteria:

1. Circulatory disease (eg pre-existing hypertension)
2. Cardiac disease/medications (e.g. angina, cardiomyopathy, B Blocker medication)
3. Pregnancy related disease (eg pre-eclampsia)
4. Diabetes pre-existing the pregnancy
5. Hyperthyroidism
6. Renal Disease
7. Closed-angle glaucoma
8. Patients on monoamine oxidase inhibitors
9. In active labour
10. Emergency caesarean section
11. Fetal abnormalities
12. Contraindications to spinal anaesthesia
13. Height >6 feet/180cm / Height <5 feet/150cm
14. Body mass index (BMI) <19 or >35

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
ST segment changes on Holter monitoring | 30 minutes pre spinal anaesthesia to 4 hours post delivery

SECONDARY OUTCOMES:
Troponin levels | 24h post delivery
Incidence of maternal low systolic blood pressure | 20 minutes post spinal and 30 minutes post delivery
Maternal cardiac output | 20 minutes post spinal and one measure at 5 minutes post delivery

CONTACTS AND LOCATIONS:
Overall Officials: Roshan Fernando, FRCA, Principal Investigator — University College London Hospital
Locations (1):
- University College London Hospital, London, United Kingdom